CLINICAL TRIAL: NCT00632944
Title: Effects of Nursing Rounds on Patients Fall Rates, Satisfaction, and Call Light Use in an In-patient Medical Surgical Unit
Brief Title: Effects of Nursing Rounds on Patients Fall Rates
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Melanie Kalman, Dr Melanie Kalman, State University of New York - Upstate Medical University
Other Study IDs: 5529
Record Dates: First submitted 2008-03-03; First posted 2008-03-11 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2008-03

CONDITIONS: Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the effects of hourly rounding on patient falls, patient satisfaction, and patient call light usage. This is a replication of research which determined that hourly rounds conducted by nursing personnel decreased patient falls and call light usage and increased patient satisfaction. The study design is quasi- experimental. One unit will be used as its own control (4S). On this unit, hourly nursing rounds will be implemented by Registered Nurses, Licensed Practical Nurses, and Nursing Assistants. A second unit, 6S, will maintain current practices and data from this unit will be used to determine if there are any hospital-wide fluctuations for fall rates, patient satisfaction, or call light usage. Data for patient falls, patient satisfaction, call light usage, and reasons for call light use will be collected on both units using fall rate reports, patient satisfaction survey data, and the call light system.

Falls among hospital patients are a persistent problem, with 2.3 to 7 falls occurring in U.S. hospitals every 1000 patient days. Approximately 30-48% percent of these falls result in injury and 5 to 10 percent of them result in serious injury. Fall related deaths occurred at a rate of 46.2 per 100,000 in 2003. Hospital falls affect both young and old patients and many of them occur when the patient is alone or involved in elimination-related activities. Falls that result in injury may lead to an extended hospitalization and increased costs. Patients who fall and sustain injury are reported to have hospital charges of more than $4,200 higher than patients who do not fall. Hourly nursing rounds have been shown to decrease falls by 52%.

Hospitalized patients often require assistance with basic self-care tasks, such as using the toilet, ambulating, and eating; they ask for assistance by using the call light. Therefore, a patient's level of satisfaction with nursing care depends principally upon the patient's perception of how well the nursing staff has been able to meet his or her needs. The call light can be a lifeline for hospitalized patients, but it can also impose considerable demands on nurses' time. Several studies have documented the unfavorable effects of patients' frequent use of call lights on the effectiveness of patient-care management on inpatient units, which may already be compromised by staffing shortages.

DETAILED DESCRIPTION:
Falls among hospital patients are a persistent problem, with 2.3 to 7 falls occurring in U.S. hospitals every 1000 patient days. Approximately 30-48% percent of these falls result in injury and 5 to 10 percent of them result in serious injury. Fall related deaths occurred at a rate of 46.2 per 100,000 in 2003. Hospital falls affect both young and old patients and many of them occur when the patient is alone or involved in elimination-related activities. Falls that result in injury may lead to an extended hospitalization and increased costs . Patients who fall and sustain injury are reported to have hospital charges of more than $4,200 higher per admission than patients who do not fall. Hourly nursing rounds have been shown to decrease falls by 52% .

Hospitalized patients often require assistance with basic self-care tasks, such as using the toilet, ambulating, and eating; they ask for assistance by using the call light. Therefore, a patient's level of satisfaction with nursing care depends principally upon the patient's perception of how well the nursing staff has been able to meet his or her needs. The call light can be a lifeline for hospitalized patients, but it can also impose considerable demands on nurses' time. Several studies have documented the unfavorable effects of patients' frequent use of call lights on the effectiveness of patient-care management on inpatient units, which may already be compromised by staffing shortages.

Current data at Crouse Hospital show that the fall rate on 4S is 5.05 per 1000 patient days, demonstrating significant opportunity for improvement. Data from the 6S shows a fall rate of 5.26 per 1000 patient days. As far as patient satisfaction, the percentage of patients who gave the 4S a 9 or 10 out of a possible score of 10 for overall rating of care was 56.29%. Likewise the number of patients who would definitely recommend Crouse Hospital to others was 56.25%. Both satisfaction questions (Core IP Key Results: I would prefer to return to X without hesitation, if care is needed and I would recommend X without hesitation to others) show significant opportunities for improvement. Preliminary call light usage gathered from the Hill Rom call light system, which is currently available only on 6S, showed 6,909 individual uses of the call light within a 4-week period. One can surmise from this number that patient issues are not being addressed in a timely manner and therefore significant opportunities for improvement exist. Only aggregate data will be collected. No subjects will be identified directly or through any identifiers.

The objectives of the study are to:

1. Correlate the effects of hourly nursing rounds, if any, to patient falls and call light use.
2. Determine if there are any changes in patient satisfaction levels

All subjects 18 years and over admitted to 4 South Irving (Oncology/OBGYN) or 6 South Irving (Orthopedic/Neurology) during the twelve month study will be included as research subjects.

Exclusion Criteria: Any patient not admitted to 4 South Irving or 6 South Irving at Crouse Hospital will be excluded from the study. Patients under the age of 18 years are not admitted to these units.

Sample sizes for the study were determined for call light usage rates, patient satisfaction scores, and fall rates. Current process averages for sample size calculations were obtained as follows: 1) fall rates from existing fall rate reports 2) patient satisfaction from Avatar surveys, and 3) call bell usage from preliminary Hill Rom system data. For all sample size calculations, α=0.05 and β=0.10 were used. Based on these calculations, the study baseline data for patient satisfaction will be calculated using Avatar patient satisfaction data from the six-month period prior to study initiation. The baseline data for falls will be collected from existing fall rate reports using the six months of data prior to study initiation. Data for these variables will continue to be collected for 6 months after the implementation of nursing rounds. For call bell usage rates the data for 2 weeks prior to rounding implementation will be collected as baseline data. Data will be collected for 4 weeks following the implementation of nursing rounds. Data for average patient age, length of stay, and severity of illness for both units will be obtained from Transition Systems, Inc. TSI, a financial data base is a type of Decision Support System. In order to get the information on a patient's age a query will be made of TSI. It will then print up average ages of a particular unit within a specified time. Measures of central tendency and spread will be calculated for these variables to compare both units. Chi-square tests, rank sum tests, and tests of means will be used to compare baseline and post-intervention demographic characteristics and reasons for call light usage on both units. Rate ratios comparing post- to pre-intervention fall rates and call rates will be calculated on both. For both fall rates and call rates, significance tests will be conducted to determine whether the rate ratios differ between the two units. The change in the proportion of patients who indicated they were satisfied with their care in each unit before and after the intervention will also be calculated and compared. The data will be analyzed using SAS®9. No data involving individual patient identifiers will be presented with the analysis. Findings from this study will potentially be used to change nursing practice at Crouse Hospital.

4-South Irving, the experimental unit, will be used as its own control. A second unit, 6S, will maintain current practices and data from this unit will be used to determine if there are any hospital-wide fluctuations for fall rates, patient satisfaction, or call light usage. Age, gender, and severity of illness of subjects on the control and experimental units will be compared. Because the patient populations differ from the experimental to control unit, the reasons why patients use the call light will be collected to verify that these two groups use the call lights for similar reasons.

The principal and co-investigators of this study will be educating all nursing personnel on both units on how to collect and document call light data 1 week prior to the start of the data collection process. Baseline call light data for the reasons why patients use the call light and number of patient calls will then be collected for 2 weeks. After baseline call light data are collected the principal and co-investigators will be educating all nursing personnel on 4 South Irving on how to round on patients. Education will last for 2 weeks and includes what questions to ask of the patient while in the room, what tasks need to be done each time they are in the room, when to round on patients, and how to document rounds. An hourly rounding toolkit purchased from the authors of the original study, which includes an educational video, will be used to assist in this education phase. Nursing leadership, which includes the nurse manager, Director of Medical-Surgical Nursing, the Chief Nursing Officer and Clinical Nurse Specialists, will be educated on techniques to ensure rounding is consistently completed by nursing personnel. The implementation of nursing rounds will begin after the two weeks of rounding education is completed.

One member of the nursing staff, including RNs, LPNs, and Nursing Assistants, will be required to perform nursing rounds every hour on 4 South Irving Patients will not be awakened if they are sleeping unless it is necessary for treatment. During nursing rounds, nursing personnel will assess pain levels using a pain-assessment scale, offer toileting assistance, assess the patient's position and position comfort, make sure the call light is within the patients reach, put the television remote control and bed light switch within the patients reach, put the bedside table next to the bed, put the tissue box and water within the patient's reach and prior to leaving the room ask "Is there anything I can do for you before I leave? I have time while I am here in the room." Nursing personnel will also tell the patient that a member of the nursing staff (name will be written on white board in room) will be back in an hour to round again. Nursing staff members are expected to complete all patient-care tasks, unless they are not authorized to dispense medication or work with IVs. Laminated pocket cards will be given to nursing staff so they are continually reminded of the actions to perform on the rounds. Patients will not be awakened to check for pain, positioning, or the need to use the bathroom; however the environmental check can be completed during rounds. Members of the nursing leadership team including the nurse manager, Director of Medical-Surgical Nursing, Chief Nursing Officer, and Clinical Nurse Specialists will be making frequent observations of staff, using rounding documentation sheets and patient interviews, to verify that rounding is occurring as expected.

Call light usage will be collected through the use of the Hill Rom call light system. Recently, Hill Rom Beds were added to 4 South. Now the two units are equipped with Hill Rom Beds and corresponding Hill Rom call lights. All call lights placed from individual patient rooms are recorded on a central server located in each nursing station. The central server can generate and print reports for all call lights used in a user specified time frame. Reports include the time a call light was placed, area it was placed from and call light response time. Reasons for call light usage will be documented by bedside nursing personnel on a standard sheet. The documentation forms will be collected every day at 7a.m. by the principal investigator or co-investigators of the study. New documentation forms will be posted daily at 7a.m. Inter-rater reliability will be performed by comparing manual call light data to the computerized call light data collected within the Hill Rom call light system. Documentation of rounding times and frequency will also be documented by nursing personnel on a standard form . This form will be collected every day at 7a.m. by either the principal investigator or co-investigator of the study. New rounding documentation forms will be posted daily. Rounding documentation forms will be used to calculate the percentage of rounds completed as expected.

On both units, baseline data collection for falls and patient satisfaction will be collected for 6 months prior to the start of nursing rounds and 6 months after the start of the implementation of nursing rounds. Fall rates will be collected through pre-existing fall rate reports and reported as falls per 1000 patient days. Patient satisfaction will be collected through pre-existing Avatar patient satisfaction surveys that are randomly sent to discharged patients. All data will be analyzed to determine if statistically significant differences in patient fall rates, satisfaction, or call light usage occurred.

A limitation in this study is that nurses from the medical surgical float pool may work on 4 South and subsequently be assigned to 6 South within the 6 month post-intervention time period. This potential movement of nurses between the control and experimental unit may influence the results on the control unit. This will be addressed by limiting the number of float pool nurses who are scheduled to work on both the experimental unit and the control unit for the six months following the education phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* All subjects 18 years and over admitted to 4 South (Oncology/OBGYN) or 6 South (Orthopedic/Neurology) at Hospital during the twelve month study will be included as research subjects.

Exclusion Criteria:

* Any patient not admitted to 4 South or 6 South at Hospital will be excluded from the study.
* Patients under the age of 18 years are not admitted to these units.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In patients on 2 units: an Oncology/OBGYN unit and an Orthopedic/Neurology unit.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Correlate the effects of hourly nursing rounds, if any, to patient falls and call light use. | 1 year

SECONDARY OUTCOMES:
Determine if there are any changes in patient satisfaction levels | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Kalman, RN PhD, Principal Investigator — SUNY UMU